CLINICAL TRIAL: NCT04083586
Title: Pattern and Frequency of Non-epileptic Involuntary Movements. Hospital-based Study
Brief Title: Pattern and Frequency of Non-epileptic Involuntary Movements
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Roaa Almoataz Abdelrazik Zohni Elsabrout, post graduate, Assiut University
Other Study IDs: frequency involuntary movement
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Involuntary Movements
MeSH Terms: conditions — Dyskinesias | interventions — Laboratories; Health Services Needs and Demand

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: All investigations; laboratory and radiological, needed for diagnosis — mri brain, ct brain, drug screening

SUMMARY:
We will perform a medical record review of all patients seen in Assiut University hospital, Egypt, to determine the frequency of movement disorders seen, disease characteristics, diagnostic evaluations.

DETAILED DESCRIPTION:
Movement disorders are conventionally divided into major categories: 1) Hyperkinetic movement disorders (also called dyskinesias) refer to excessive, often repetitive, involuntary movements that intrude into the normal flow of motor activity. This category includes chorea, dystonia, myoclonus, stereotypies, tics, and tremor. 2) Hypokinetic movement 3) Ataxia.

Hyperkinetic movements any unwanted excess movement. Together with hypertonia (abnormally increased resistance to externally imposed movement) and negative signs (insufficient muscle activity or insufficient control of muscle activity).

Tremor: Tremor is a rhythmic back-and-forth or oscillating purposeless involuntary movement about a joint axis. Tremor occurs at rest (the pill-rolling tremor of Parkinsonism). Postural tremor (the fine tremor of hyperthyroidism), Action tremor (intention tremor) occurs near the end of a goal-directed movement.

Chorea : is a series of brief, jerky, explosive ongoing random-appearing sequence of one or more discrete involuntary movements, or "fidgeting; there are different causes of chorea, Sydenham's chorea. Lesions in the sub thalamic nucleus. Encephalitis with diffuse gray-matter. Motor impersistence is a common association.

Athetosis is a slow, continuous, writhing, sinuous movement, especially marked in the digits and extremities, prevents maintenance of a stable posture.

Myoclonus consists of sequence of repeated, often non-rhythmic sudden brief twitches or jerks or involuntary contraction or relaxation of one or more muscles as seen in metabolic encephalopathies such as uremic encephalopathy. It can be categorized as "action myoclonus", "postural myoclonus", or "rest myoclonus" based on the condition when it is observed Asterixis :is an intermittency of sustained posture, illustrated by "flapping" of the hands when the arms are outstretched and wrists dorsiflexed, as in hepatic encephalopathy.

Stereotypies are repetitive, simple movements that can be voluntarily suppressed. Stereotypies do not necessarily hold the person's attention.

Tics are repeated, individually recognizable, intermittent movements that are almost always briefly suppressible and are usually associated with awareness of an urge to perform the movement.

Dystonia: a movement disorder in which involuntary sustained or intermittent muscle contractions cause twisting and repetitive movements, abnormal postures, or both. Dystonic postures are often triggered by attempts at voluntary movement or voluntary posture, as may occur in task-specific dystonia.

Hypokinetic movements: include bradykinesia (slowness of movement) and hypokinesia (poverty of movement, and movements that are smaller than intended), but also crucially and fundamentally the progressive fatiguing and decrement of repetitive alternating movements seen during finger or foot tapping. The best known cause and example is Parkinson's disease.

Ataxia: Ataxia is a degenerative disorder affecting the brain, brainstem or spinal cord. This can result in clumsiness, inaccuracy, instability, imbalance, tremor or a lack of coordination while performing voluntary movements. Ataxia also can affect speech and movement of the eyes.

Previous epidemiological studies in Egypt showed that the Overall the recorded Crude Prevalence Rate (CPR) of Parkinson's disease in Egypt was varied in different governorates and ranged from 53 to 557/105 inhabitants Another study was planned to estimate the prevalence and to study the aetiological factors of chorea, dystonia, athetosis and hemiballismus in Assiut. The prevalence rate for rheumatic chorea was 62/100,000 population, whereas Huntington's chorea had a prevalence rate of 21/100,000. The other two common types of chorea were reported with prevalence rates of 12/100,000 for the encephalitic type and 17/100,000 for the atherosclerotic type. No single case of generalized dystonia was recorded and all cases were of the focal type of dystonia with a prevalence rate of 26/100,000 population, but there's no available data about other movement disorders in Egypt

ELIGIBILITY:
Inclusion Criteria:

* Patients with movement disorders attending Assiut University neurology outpatient clinic and internal department, from Jan 2020 to Jan 2021.

Exclusion Criteria:

* 1) involuntary movements epileptic in origin 2) refusal of patient to give consent to join the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with movement disorders attending Assiut University neurology outpatient clinic and internal department, from Jan 2020 to Jan 2021.
  sample size: regarding previously estimated prevalence in (kwon KY et al,2019), was 292, so our sample size as calculated: Sample Size(n) for Various Confidence Levels ________________________________________ Confidence Level(%) Sample Size 95% 167 80% 106 90% 141 97% 181 99% 203 99.9% 231 99.99% 245
  ________________________________________ Equation Sample size n = [DEFF*Np(1-p)]/ [(d2/Z21-α/2*(N-1)+p*(1-p)]
  Results from OpenEpi, Version 3, open source calculator--SSPropor
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
•Detect pattern and clinical characteristics of patients with different forms of movement disorders attending Assiut University neurology outpatient clinic and internal department as parkinson's disease | from Dec15th 2019 to June15th 2020.
  Using MDS- Unified Parkinson's Disease Rating Scale (UPDRS) (Goetz et al., 2008) for PD. (parts 3) III: Motor Examination, The investigator should "rate what you see.concurrent medical problems and orthopedic problems may interfere with individual items in the motor examination. In situations where it is absolutely impossible to test use the notation "UR" for Unable to Rate. Otherwise, rate the performance of each task as the patient performs in the context of co-morbidities.Do higher values represent a worse outcome
•Detect pattern and clinical characteristics of patients with different forms of movement disorders attending Assiut University neurology outpatient clinic and internal department as dystonia | from Dec15th 2019 to June15th 2020.
  using Fahn-Marsden rating scale (FMRS), for dystonia. The FMDRS is composed of two clinician-rated subscales: a movement subscale, based on patient examination, and a disability subscale, based on the patient's report of disability in activities of daily living.The movement subscale rates dystonia severity and provoking factors in nine body areas, All items have a 5-point score. The provoking factor rates the relation of dystonia to action, from 0 (no dystonia at rest or with action) to 4 (dystonia at rest).The maximal total FMDRS score is 120. The disability subscale is composed of 7 items for activities of daily living,providing a maximum disability sub- score of 30. Do higher values represent a worse outcome
•Detect pattern and clinical characteristics of patients with different forms of movement disorders attending Assiut University neurology outpatient clinic and internal department as essential tremors | from Dec15th 2019 to June15th 2020.
  Using • Tremor assessment form (TAF) for tremor: A questionnaire related to hand tremor consisting of 12 items was prospectively applied to patients with PD or ET in three movement-disorder clinics. Each question was analyzed, and a query-based scoring system was evaluated for differentiating hand tremors between PD and ET

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy El-Tallawy, professor, Study Chair — Professor of Neurology Faculty of Medicine, Assiut University; Ali Shalash, professor, Study Director — Professor of Neurology Faculty of Medicine, Ain Shams University; mohamed abdelhameed, assist prof, Study Director — Assistant professor of Neurology Faculty of Medicine, Assiut University; roaa elsabrout, postgraduate, Principal Investigator — Resident at neuropsychiatry department Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Sanger TD, Chen D, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Taskforce on Childhood Motor Disorders. Definition and classification of negative motor signs in childhood. Pediatrics. 2006 Nov;118(5):2159-67. doi: 10.1542/peds.2005-3016. PMID 17079590
- [Background] Swedo SE. Sydenham's chorea. A model for childhood autoimmune neuropsychiatric disorders. JAMA. 1994 Dec 14;272(22):1788-91. doi: 10.1001/jama.272.22.1788. No abstract available. PMID 7661914
- [Background] Benabid AL, Benazzouz A, Limousin P, Koudsie A, Krack P, Piallat B, Pollak P. Dyskinesias and the subthalamic nucleus. Ann Neurol. 2000 Apr;47(4 Suppl 1):S189-92. PMID 10762147
- [Background] Janavs JL, Aminoff MJ. Dystonia and chorea in acquired systemic disorders. J Neurol Neurosurg Psychiatry. 1998 Oct;65(4):436-45. doi: 10.1136/jnnp.65.4.436. PMID 9771763
- [Background] Cardoso F, Eduardo C, Silva AP, Mota CC. Chorea in fifty consecutive patients with rheumatic fever. Mov Disord. 1997 Sep;12(5):701-3. doi: 10.1002/mds.870120512. PMID 9380051
- [Background] Morris JG, Jankelowitz SK, Fung VS, Clouston PD, Hayes MW, Grattan-Smith P. Athetosis I: historical considerations. Mov Disord. 2002 Nov;17(6):1278-80. doi: 10.1002/mds.10267. No abstract available. PMID 12465068
- [Background] Caviness JN, Brown P. Myoclonus: current concepts and recent advances. Lancet Neurol. 2004 Oct;3(10):598-607. doi: 10.1016/S1474-4422(04)00880-4. PMID 15380156
- [Background] Kennedy CH, Meyer KA, Knowles T, Shukla S. Analyzing the multiple functions of stereotypical behavior for students with autism: implications for assessment and treatment. J Appl Behav Anal. 2000 Winter;33(4):559-71. doi: 10.1901/jaba.2000.33-559. PMID 11214031
- [Background] Swedo SE, Leonard HL, Garvey M, Mittleman B, Allen AJ, Perlmutter S, Lougee L, Dow S, Zamkoff J, Dubbert BK. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections: clinical description of the first 50 cases. Am J Psychiatry. 1998 Feb;155(2):264-71. doi: 10.1176/ajp.155.2.264. PMID 9464208
- [Background] Meierkord H, Fish DR, Smith SJ, Scott CA, Shorvon SD, Marsden CD. Is nocturnal paroxysmal dystonia a form of frontal lobe epilepsy? Mov Disord. 1992;7(1):38-42. doi: 10.1002/mds.870070107. PMID 1557065
- [Background] El-Tallawy HN, Farghaly WM, Shehata GA, Rageh TA, Hakeem NM, Hamed MA, Badry R. Prevalence of Parkinson's disease and other types of Parkinsonism in Al Kharga district, Egypt. Neuropsychiatr Dis Treat. 2013;9:1821-6. doi: 10.2147/NDT.S48318. Epub 2013 Nov 26. PMID 24379673